CLINICAL TRIAL: NCT07008482
Title: Effects of Music on Preoperative Anxiety in Patients With Femoral Fractures Scheduled for Surgical Intervention: A Randomized Controlled Study
Brief Title: Effects of Music on Preoperative Anxiety in Patients With Femoral Fractures Undergoing Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Principal Investigator, Massimo Guasconi, RN, MSN, Azienda Unita Sanitaria Locale di Piacenza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SINFEMIA
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Pain; Surgery; Femoral Fractures; Music Therapy
Keywords: NURSING; MUSICTHERAPY; ANXIETY; PAIN
MeSH Terms: conditions — Anxiety Disorders; Pain; Femoral Fractures

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Data processing will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MUSIC THERAPY (Experimental)
  Interventions: Other: Music intervention
- NO MUSICTHERAPY (No Intervention)

INTERVENTIONS:
Other: Music intervention — patient enrolment, administration of the APAIS and NRS scales (T0), administration of the standard music therapy/assistance intervention (20 minutes duration), re-evaluation with re-administration of the APAIS and NRS scales (T1) and completion of the CRF. The administration will take place at the patient's bedside, respecting the privacy and confidentiality of the subjects involved, guaranteeing absolute tranquillity, also with the help of dividers to avoid distractions and interruptions.
  Arms: MUSIC THERAPY

SUMMARY:
This randomized controlled trial (RCT) investigates the effectiveness of music therapy in reducing preoperative anxiety among elderly patients with femoral fractures. Preoperative anxiety is known to worsen physiological stability, increase pain perception, and negatively impact recovery, yet specific evidence on non-pharmacological interventions like music therapy in the orthogeriatric setting is lacking.

The study will enroll 154 adult patients admitted to the Orthogeriatrics Unit for elective femoral fracture surgery. Participants will be randomly assigned to receive either a 20-minute session of music therapy or standard care. Anxiety will be measured using the APAIS scale, and pain will be assessed with the NRS scale, both before and after the intervention.

The trial is designed as a blinded, prospective RCT, with data collected and managed under current privacy regulations. By generating robust data on this low-cost, safe intervention, the study aims to improve preoperative management and patient outcomes in orthopedic surgical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, 18 years of age or older
* Patients with femur fracture who are candidates for surgery
* Able to provide informed consent.

Exclusion Criteria:

* Patients with a diagnosis of hearing loss
* Patients diagnosed with cognitive or psychiatric disorders
* Patients undergoing emergency/emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference between the Amsterdam Preoperative Anxiety and Information Scale (APAIS) at T0 and T1 | Baseline and 20 minutes after baseline
  Difference in preoperative anxiety level after 20 minutes and baseline evaluated by APAIS scores between T0 and T1. The APAIS consists of six questions, with each question rated on a 5-point Likert scale (1=not at all, 5=extremely), and has a minimum score of 6 and a maximum score of 30. Higher APAIS scores indicate a worse outcome with higher levels of anxiety and a greater desire for information.

IPD SHARING:
Plan to Share IPD: Undecided